CLINICAL TRIAL: NCT01680900
Title: Vilazodone for Menopausal Hot Flashes: A Proof in Principle Study
Brief Title: Vilazodone for Menopausal Hot Flashes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Ellen Freeman, Research Profesor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 816164
Record Dates: First submitted 2012-08-28; First posted 2012-09-07 (Estimated); Results first posted 2015-01-14 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2014-12

CONDITIONS: Hot Flushes
Keywords: menopause; hot flashes; vilazodone
MeSH Terms: conditions — Hot Flashes | interventions — Vilazodone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- experimental 1 (Experimental): vilazodone (viibryd). 20 mg or 40 mg/day for 8 weeks
  Interventions: Drug: vilazodone
- placebo capsules (sugar pill) (Placebo Comparator): Placebo capsules matched to the drug dose for 8 weeks
  Interventions: Drug: placebo capsules

INTERVENTIONS:
Drug: vilazodone — capsules once/day for 8 weeks. Dose starts at 10 mg for 7 days, increases to 20 mg/day for 7 days, increases to 40 mg/day at week 3 of unimproved.
  Other Names: viibryd
  Arms: experimental 1
Drug: placebo capsules — placebo capsules matched to drug capsules.
  Arms: placebo capsules (sugar pill)

SUMMARY:
This is a pilot study to determine proof in principle that vilazodone, a selective serotonin reuptake inhibitor and 5HT1a agonist, reduces the frequency and severity of menopausal hot flashes relative to placebo. A secondary aim is to evaluate improvement in menopause-related quality of life.

DETAILED DESCRIPTION:
This is a proposal to conduct a small clinical trial for proof in principle that vilazodone reduces the frequency and severity of menopausal hot flashes. An additional exploratory aim is to identify improvement in menopause-related quality of life. Healthy, perimenopausal women ages 45-60 with an average of 4 or more moderate or severe hot flashes/night sweats per day for 3 screening weeks will be randomized to 8 weeks of treatment in a 2:1 ratio of vilazodone or matching placebo pills. Flexible dosing of vilazodone will start at 10 mg once/day for 7 days, increase to 20 mg/day for 1 more week and increase to 40 mg once/day at week 3 if unimproved. The primary outcome assessments are the frequency and severity of hot flashes at week 4 and week 8 as assessed by prospective daily diaries (using 7-day mean scores from the daily diaries). The secondary outcome is clinical improvement, defined as hot flash frequency >=50% decrease from baseline. Treatment-emergent adverse events will be monitored and patient ratings of tolerability will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 45-60 years
* Amenorrhea for 60 days or more or postmenopausal or bi-lateral oophorectomy.
* 4 or more moderate or severe hot flashes or night sweats per 24 hour period (28/week) as recorded on daily diaries in 3 screening weeks.
* Hot flashes/night sweats rated as moderate to severe and/or bothersome (moderately to a lot) on 4 or more days/nights in each screen week.
* In general good health.
* Signed informed consent.

Exclusion Criteria:

* Psychotropic medications currently or within the last 30 days.
* Current use of hormonal medications such as hormone therapy or hormonal contraception or any treatment for hot flashes (Prescription, over-the-counter or herbal).
* Drug or alcohol abuse in the past year.
* Lifetime diagnosis of psychosis or bipolar disorder.
* Suicide attempt in the past 3 years or any current suicidal ideation.
* Current major depression.
* Not using a medically approved, non-hormonal method of birth control if sexually active and not postmenopausal (12 or more months since last menstrual period or bi-lateral oophorectomy).
* Pregnancy, intending pregnancy or breast feeding.
* Any severe of unstable medical illness, e.g., breast or ovarian cancer, seizure disorders, etc.
* Current participation in another intervention study.
* Inability or unwillingness to complete study procedures.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen W Freeman, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Dept OB/GYN, Mudd Professorship Suite, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental 1 | Placebo Capsules (Sugar Pill)
Started | 24 | 12
Completed | 20 | 11
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental 1 | Placebo Capsules (Sugar Pill) | Total
Number analyzed (Participants) | 24 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] — self-reported age in years
  years | 51.5 (3.7) | 52.7 (4.2) | 51.9 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 12 | 36
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: Daily Diary Ratings of Frequency of Hot Flashes
Description: Hot flash frequency and severity will be recorded daily in the am and pm on a scale of 0 (none) to 3 (severe). The frequency of hot flashes was the number reported.
Time Frame: Week 8.
Population: all participants randomized to treatment
Measure: Mean (95% Confidence Interval); unit: number of hot flashes
Arm/Group | Experimental 1 | Placebo Capsules (Sugar Pill)
Number analyzed (Participants) | 24 | 12
number of hot flashes | 3.65 [2.57 to 4.73] | 4.71 [3.61 to 5.80]
Statistical Analysis 1: Comparison: Experimental 1 vs Placebo Capsules (Sugar Pill); Test type: Superiority or Other; p = 0.05, Regression, Linear; Mean Difference (Final Values) = -1.06, 95% CI 2-sided [-2.60 to -0.48]

2. Secondary Outcome: Percent of Patients With >=50% Reduction in Moderate to Severe Hot Flashes
Description: Percent of patients with n >=50% reduction in frequency of moderate to severe hot flashes calculated from daily diaries
Time Frame: Percent change from baseline at Week 8
Population: all participants with at least one treatment response
Measure: Number; unit: percentage of participants
Arm/Group | Experimental 1 | Placebo Capsules (Sugar Pill)
Number analyzed (Participants) | 24 | 12
percentage of participants | 65 | 83
Statistical Analysis 1: Comparison: Experimental 1 vs Placebo Capsules (Sugar Pill); Test type: Superiority or Other; p < 0.05, Chi-squared

3. Secondary Outcome: Menopause-related Quality of Life (MENQOL)
Description: The MENQOL is a validated measure to assess the presence and bother of menopausal symptoms. This will be exploratory. Each of 29 items is rated on a scale of 0 to 6 (extremely bothersome). The items are divided into 4 subscales. The item scores are summed in each subscale and means are computed for the 4 subscales. The total score is the sum of the mean subscale scores. Higher scores are more symptomatic.
Time Frame: Week 8
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Experimental 1 | Placebo Capsules (Sugar Pill)
Number analyzed (Participants) | 24 | 12
units on a scale | 1.89 [1.55 to 2.24] | 2.08 [1.63 to 2.53]
Statistical Analysis 1: Comparison: Experimental 1 vs Placebo Capsules (Sugar Pill); Test type: Superiority or Other; p < 0.05, Regression, Linear; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.75 to -0.08]

4. Other Pre Specified Outcome: Number of Participants With Adverse Events
Description: A 17 item checklist of general adverse and withdrawal symptoms. It will be used at baseline and Week 12. Adverse events will be obtained by subject report at Week 4 and Week 8.
Time Frame: Baseline and Week 12
Measure: Number; unit: participants
Arm/Group | Experimental 1 | Placebo Capsules (Sugar Pill)
Number analyzed (Participants) | 24 | 12
participants | 17 | 6

5. Other Pre Specified Outcome: Percentage of Participants That Were Satisfied or Very Satisfied
Description: Patient global rating of satisfaction with medication reported on a scale of 0 to 5 (very satisfied).
Time Frame: Week 8
Population: all participants with at least one treatment response.
Measure: Number; unit: percentage of participants
Arm/Group | Experimental 1 | Placebo Capsules (Sugar Pill)
Number analyzed (Participants) | 24 | 12
percentage of participants | 65 | 75

6. Other Pre Specified Outcome: Sheehan Global Ratings of Symptom (Hot Flash)Interference
Description: Global ratings on a 10-point scale of the degree that symptoms interfere overall, with work, social activities and family life.
Time Frame: Change from Baseline at Week 8
Reporting Status: Not Posted

7. Primary Outcome: Daily Diary Ratings of Severity of Hot Flashes
Description: Hot flash severity will be recorded daily in the am and pm on a scale of 0 (none) to 3 (severe). The frequency of hot flashes was the number reported. The severity of hot flashes was rated on a scale of 0 (none) to 3 (severe). 7-day averages were calculated for baseline, week 4 and week 8 and a mean daily score was obtained for analysis. Baseline values were the means of the first 2 screen weeks. Possible range of the severity scale for the daily mean was 0 (none) to 3 (severe).
Time Frame: Week 8.
Population: all participants randomized to treatment
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Experimental 1 | Placebo Capsules (Sugar Pill)
Number analyzed (Participants) | 24 | 12
units on a scale | 1.17 [1.05 to 1.80] | 1.39 [1.02 to 1.76]
Statistical Analysis 1: Comparison: Experimental 1 vs Placebo Capsules (Sugar Pill); Test type: Superiority or Other; p = 0.05, Regression, Linear; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.74 to -0.21]

ADVERSE EVENTS:
Arm/Group | Experimental 1 | Placebo Capsules (Sugar Pill)
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/12
Other Adverse Events (participants affected / at risk) | 17/24 | 6/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental 1 (N=24) | Placebo Capsules (Sugar Pill) (N=12)
diarrhea (Gastrointestinal disorders) | 9 | 0
nausea (Gastrointestinal disorders) | 7 | 0
headache (Nervous system disorders) | 4 | 2
dry mouth (Nervous system disorders) | 4 | 3
dehydration (Gastrointestinal disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No